CLINICAL TRIAL: NCT05737433
Title: An Open Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Rencofilstat in Healthy Male Subjects
Brief Title: Single Dose ADME Study of [14C]-Rencofilstat in Healthy Male Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hepion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEPA-CRV431-105
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: NASH With Fibrosis
Keywords: Nonalcoholic Steatohepatitis; NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — CRV-431

STUDY DESIGN:
Intervention Model Description: open label, non-randomized, single period, and single dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]-RCF 225mg (Experimental): [14C]-rencofilstat, 225mg oral dose, self-micro-emulsifying drug delivery system, single dose
  Interventions: Drug: [14C]-rencofilstat 225mg

INTERVENTIONS:
Drug: [14C]-rencofilstat 225mg — radio-labelled 225mg oral dose of rencofilstat
  Other Names: CRV431

SUMMARY:
This is a single-center, single-period, single-dose, open-label, non-randomized study to assess the mass balance recovery, metabolite profile and metabolite identification of 14C- labelled rencofilstat ([14C] CRV431). It is planned to enroll 6 healthy male subjects in a single group. Each subject will receive a single 225 mg oral dose of [14C] CRV431 self-micro emulsifying drug delivery system (SMEDDS) oral emulsion.

DETAILED DESCRIPTION:
This is a single center, open-label, non-randomized, single period, single dose study in healthy male subjects designed to assess the mass balance recovery, pharmacokinetics (PK), metabolite profile and metabolite identification of rencofilstat. It is planned to enroll a single cohort of 6 subjects. All subjects will receive a single 225 mg oral dose of [14C]-rencofilstat, as a SMEDDS oral emulsion in the fasted state.

Subjects will undergo preliminary screening procedures for the study at the screening visit (Day -28 to Day -2). Subjects will be admitted in the evening on the day before dosing (Day-1).

Whole blood, plasma, urine and feces samples will be collected at regular intervals for PK analysis, total radioactivity analysis, metabolite profiling, mass balance and safety as applicable, from pre-dose to discharge from the clinical unit. Urine and feces samples may be collected at return visits or home visits if mass balance criteria have not been met by a subject.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Aged 30 to 65 years inclusive at the time of signing informed consent
3. Body mass index (BMI) of 18.0 to 35.0 kg/m2 as measured at screening
4. Must be willing and able to communicate and participate in the whole study
5. Must have regular bowel movements (ie average stool production of ≥1 and ≤3 stools per day)
6. Must provide written informed consent
7. Must agree to adhere to the contraception requirements

Exclusion Criteria:

1. Subjects who have received any investigational treatment in a clinical research study within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer
2. Subjects who are, or are immediate family members of, a study site or sponsor employee
3. Evidence or history of current SARS-CoV-2 infection within 4 weeks prior to study drug administration
4. History of any drug or alcohol abuse in the past 2 years prior to screening
5. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
6. A confirmed positive alcohol breath test at screening or admission
7. Current smokers and those who have smoked within the last 12 months prior to screening
8. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
9. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months prior to screening
10. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
11. Subjects who do not have suitable veins for multiple venipunctures/cannulation as assessed by the investigator or delegate at screening
12. Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator. Subjects known to have Gilbert's syndrome are excluded
13. Confirmed positive drugs of abuse test result
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
15. Evidence of renal impairment at screening, as indicated by an estimated eGFR of <60 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration equation
16. History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, malabsorptive, neurological or psychiatric disorder, as judged by the investigator
17. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
18. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
19. Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
20. Subjects who have taken known strong or moderate CYP3A4 inducers in the 30 days before IMP administration
21. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day) in the 14 days before study drug administration. Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no pharmacodynamic activity is expected by the time of dosing with study drug; and if the use of medication does not jeopardize the safety of the trial subject; and if the use of medication is not considered to interfere with the objectives of the study
22. Subjects who have had a COVID-19 vaccine 7 days before dosing

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MD, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After subjects consented for study, they went through the screening process. Subjects that qualified for study were assigned to the single treatment arm.
Period: Overall Study
Arm/Group | [14C]-RCF 225mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline population contains 6 six subjects. The same subjects are in the pharmacokinetic population and safety population.
Arm/Group | [14C]-RCF 225mg
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 6
% of [14C]-RCF recovered [Number; unit: %] | 0

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Mass Balance Recovery After a Single Oral Dose of [14C]-Rencofilstat
Description: Cumulative percentage of total radioactivity recovered after a single oral dose of [14C]-rencofilstat.
Time Frame: 22 Days
Population: Mass balance population
Measure: Number; unit: percentage of total radioactivity
Arm/Group | [14C]-RCF 225mg
Number analyzed (Participants) | 6
percentage of total radioactivity | 91

ADVERSE EVENTS:
Time Frame: 63 days, screening period to on study last visit.
Arm/Group | [14C]-RCF 225mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]-RCF 225mg (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT05737433/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT05737433/SAP_001.pdf